CLINICAL TRIAL: NCT03054623
Title: Prospective Hemodynamic Assessment of Distal Revascularization Interval Ligation
Brief Title: Hemodynamic Assessment of Distal Revascularization Interval Ligation
Acronym: DRIL
Status: Terminated | Type: Observational
Why Stopped: PI Left Institution
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: DRIL
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Steal Syndrome; Chronic Kidney Diseases; Arterio-Venous Fistula
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DRIL procedure: Adult (>18 yo) patients with chronic kidney disease with functioning antecubital-based arteriovenous fistulae and evidence of ischemic steal symptoms
  Interventions: Procedure: DRIL procedure

INTERVENTIONS:
Procedure: DRIL procedure — The DRIL procedure involves creation of a bypass from an arterial inflow site (usually mid brachial artery) proximal to the fistula inflow, to the bifurcation of the brachial artery distal to the fistula, with ligation of the intervening native vessel, thus restoring distal flow while preserving flow through the fistula.

SUMMARY:
Our study seeks to define the effect of each component of the distal revascularization interval ligation (DRIL) procedure on the in vivo distal blood pressure of patients with ischemic steal, and to determine whether the interval ligation component of the DRIL procedure is necessary or not.

DETAILED DESCRIPTION:
This study will involve identification of patients with ischemic steal who are deemed candidates for distal revascularization with interval ligation (DRIL), followed by prospective data collection of intraoperative noninvasive data at key points in the operation.

After informed consent, chart review will be performed to identify patient characteristics as well as details of their presentation of steal syndrome, including symptomatology, duration, characteristics of contributory arteriovenous access, and preoperative data including upper extremity/forearm pressures, fistula flow data, and finger pressures with and without fistula compression.

Patients will have noninvasive intraoperative measurement of bilateral forearm blood pressure measurements using automated blood pressure cuffs within sterile bands on the operative side as well as the contralateral ("control") side. Automated blood pressure measurements will then be performed at four time points in the operation, simultaneously on both arms (operative versus control):

1. After surgical exposure but before any intervention has been performed,
2. After clamping of the brachial artery after dissection and control of the vessel to assess for the effect of interval ligation (IL) alone on the forearm blood pressure.
3. After performance of the distal revascularization (DR) but BEFORE interval ligation of the brachial artery.
4. After completion of the procedure, including both distal revascularization AND interval ligation (DRIL).

The performance of blood pressure measurements will not alter the performance of the operation, nor will this have any influence on intraoperative decision-making. Intraoperative patient positioning and set-up will be unaffected by the addition of a distal forearm blood pressure cuff for data acquisition. Neither the pre-operative selection or post-operative care will be influenced by participation in this study, nor by the data acquired. It should be noted that this technique is intermittently used as standard of care when needed in current practice.

Patients will be assessed for symptom improvement and DRIL patency at their standard 14 day, 3 month, 6 month, 9 month and 1 year follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* >18 yo patients with CKD with a functioning antecubital-based arteriovenous fistula and evidence of ischemic steal as defined above

Exclusion Criteria:

* Patients identified as undergoing "prophylactic" or "preemptive" DRIL procedure at the time of fistula/graft creation (ie, do not have documented steal at present)
* Patients unable to provide informed consent, life expectance of less than one year
* Inability to reliably or accurately measure contralateral blood pressures due to heavily calcified vessels documented preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 yo) patients with chronic kidney disease with functioning antecubital-based arteriovenous fistulae and evidence of ischemic steal symptoms
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-08-11 (Actual)

PRIMARY OUTCOMES:
Difference in forearm pressures | one year

SECONDARY OUTCOMES:
Proportion of interval ligation procedures | one year

CONTACTS AND LOCATIONS:
Overall Officials: Karl Illig, MD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida South Tampa Campus, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zanow J, Krueger U, Reddemann P, Scholz H. Experimental study of hemodynamics in procedures to treat access-related ischemia. J Vasc Surg. 2008 Dec;48(6):1559-65. doi: 10.1016/j.jvs.2008.06.040. Epub 2008 Sep 4. PMID 18771888
- [Background] Aimaq R, Katz SG. Using distal revascularization with interval ligation as the primary treatment of hand ischemia after dialysis access creation. J Vasc Surg. 2013 Apr;57(4):1073-8; discussion 1078. doi: 10.1016/j.jvs.2012.10.085. Epub 2013 Jan 29. PMID 23375137
- [Background] Leake AE, Winger DG, Leers SA, Gupta N, Dillavou ED. Management and outcomes of dialysis access-associated steal syndrome. J Vasc Surg. 2015 Mar;61(3):754-60. doi: 10.1016/j.jvs.2014.10.038. Epub 2014 Dec 9. PMID 25499703
- [Result] Illig KA, Surowiec S, Shortell CK, Davies MG, Rhodes JM, Green RM. Hemodynamics of distal revascularization-interval ligation. Ann Vasc Surg. 2005 Mar;19(2):199-207. doi: 10.1007/s10016-004-0162-y. PMID 15770367
- [Result] Varble N, Day S, Phillips D, Mix D, Schwarz K, Illig KA, Chandra A. In vitro hemodynamic model of the arm arteriovenous circulation to study hemodynamics of native arteriovenous fistula and the distal revascularization and interval ligation procedure. J Vasc Surg. 2014 May;59(5):1410-7. doi: 10.1016/j.jvs.2013.04.055. Epub 2013 Jul 9. PMID 23845661